CLINICAL TRIAL: NCT06648928
Title: Clinician Supported Mobile App to Reduce Mental Health Symptoms Among World Trade Center Responders in Florida
Acronym: PTSDCoach911
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1 U01OH012773-01-00; U01OH012773 (NIH)
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: PTSD Symptoms; Anxiety Symptoms; Depression Symptoms; Sleep Disturbance
Keywords: First responders; World Trade Center; Randomized Clinical Trial; Mental Health; Telehealth; Latinx
MeSH Terms: conditions — Anxiety Disorders; Depression; Parasomnias; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinician Supported PTSD Coach (Experimental): PTSD Coach application combined with remotely delivered clinician support, focusing on app use, symptom monitoring, and management strategies.
  Interventions: Behavioral: Clinician Supported PTSD Coach
- Self Managed PTSD Coach application (Active Comparator): Participant remotely receives basic instructions on using the PTSD Coach application but receives no further clinician support
  Interventions: Behavioral: Self Managed PTSD Coach
- Wait list control (No Intervention): No intervention until after the follow-up assessment when they have a choice of receiving either CS PTSD Coach or SM PTSD Coach.

INTERVENTIONS:
Behavioral: Clinician Supported PTSD Coach — Combines self-managed PTSD Coach application with four 20-30 minute sessions delivered by a clinician. The app includes modules on learning about PTSD, self-assessment, symptom management, and finding support.
  Arms: Clinician Supported PTSD Coach
Behavioral: Self Managed PTSD Coach — A widely available mobile application designed to help individuals manage PTSD symptoms available in English and Spanish.
  Arms: Self Managed PTSD Coach application

SUMMARY:
This study focuses on the mental health challenges faced by the World Trade Center's (WTC) General Responders due to the severe psychological trauma from the WTC collapse. PTSD and depression are among the top mental health conditions affecting these responders. Many members of the WTC Health Program (WTCHP) have relocated to Florida, making up nearly six percent of the cohort. Furthermore, many identify as Latinx, highlighting the need for services in their preferred language to promote health equity. Studies have shown that remotely-delivered, clinician-supported applications (apps) can reduce adverse MH symptoms.

PTSD Coach was developed by the Veteran's Administration as a self-managed mobile app and is available at no cost for Android and Apple devices. The primary focus of PTSD Coach is on managing PTSD symptoms. The app offers coping tools such as relaxation exercises and calming self-talk and effective sleep hygiene practices when needed. A recent review evaluated the self-managed PTSD Coach app and found it to be feasible, acceptable, and effective in reducing PTSD symptoms.

Clinician-Supported PTSD Coach was developed as a brief intervention for Veterans who were unlikely to use a mobile app on their own. Clinician Supported PTSD Coach combines PTSD Coach mobile app with four remotely-delivered 20-30 minute sessions over 8 weeks with a clinician. Studies with Veterans have reported significant reductions in PTSD and depression symptoms, treatment satisfaction and more treatment sessions attended, when compared with typical mental health care. While promising, none of these studies included WTC General Responders or focused on Latinx populations.

Given the promise of these interventions, and the need to provide support for geographically dispersed General Responders in Florida, this study aims to evaluate the feasibility, acceptability, and effectiveness of Clinician Supported PTSD Coach in reducing symptoms of PTSD, depression, anxiety, and sleep disturbances among English and Spanish-speaking WTC General Responders. Participants will be randomly assigned to one of three conditions:

1. Clinician-Supported PTSD Coach
2. Self-Managed PTSD Coach
3. Waitlist Control (no treatment until after follow-up)

Assessments will be conducted at the end of treatment (8 weeks) and at follow-up (12 weeks). The study will measure reductions in PTSD, depression, anxiety, and sleep disturbances at 8 weeks and 12 weeks. It is expected that both Clinician Supported PTSD Coach and Self-Managed PTSD Coach will reduce symptoms, with Clinician Supported PTSD Coach showing larger reductions. In addition, to assess feasibility and acceptability, the study will assess engagement, satisfaction, and barriers in both PTSD Coach app conditions.

This project aims to fill a significant gap in evidence-based mental health treatments for WTC General Responders. It responds to the WTCHP Scientific Technical Advisory Committee's call for more research on mental health interventions and addresses the critical shortage of rigorously tested app-based remote interventions for dispersed General Responders with PTSD. The study also focuses on Spanish-speaking Latinx General Responders, a group that has not been specifically targeted in previous interventions. The study's findings could lead to the development of readily deployable interventions nationally to meet the mental health needs of WTC responders and survivors, providing a valuable resource for treatment researchers and health care providers.

DETAILED DESCRIPTION:
INTRODUCTION, BACKGROUND AND SIGNIFICANCE. The September 11, 2001 terrorist attacks on the World Trade Center (WTC) have had long-lasting impacts on the mental health of the responders involved in the rescue and recovery efforts. The World Trade Center Health Program (WTCHP) was established to monitor and treat health conditions related to the WTC disaster. This study aims to address the mental health (MH) treatment needs of WTC responders, particularly those who have relocated to Florida after retirement, therefore representing the older group of the WTCHP population and with a higher percentage of Latinos. The research focuses on evaluating the effectiveness of a clinician-supported mobile application, Clinician Supported (CS) PTSD Coach, in reducing symptoms of Post-Traumatic Stress Disorder (PTSD), depression, anxiety, and sleep disturbances among these responders. Additionally, the study emphasizes the inclusion of Spanish-speaking Latinx responders to advance health equity through the use of a Spanish version of the mobile application and Spanish adaptation of the intervention manual.

Background. Since its inception in 2011, the WTCHP, funded by the CDC/NIOSH, has been responsible for the health monitoring and treatment of over 120,000 members. These members include responders and survivors who have been diagnosed with various WTC-related health conditions. Among these conditions, mental health issues such as PTSD, anxiety, depression, substance abuse, and sleep disturbances are prevalent. Research on the WTC cohort has documented that PTSD is the most commonly certified psychiatric condition, with a prevalence ranging from 3.8% to 29.6%. Other mental health conditions include anxiety, depression, substance abuse, and sleep disturbances. Despite the chronic nature of these conditions, there is a significant gap in controlled studies on effective treatments. Most of the existing treatments have been in-person and focused on highly exposed individuals. There have been very few controlled studies, and no studies have been conducted with app-based remote interventions to serve the large number of General Responders (GRs) with full or subthreshold PTSD. Furthermore, interventions with a focus on Spanish-speaking Latinx GRs have not been conducted. This study aims to fill this gap by proposing a novel approach using a clinician-supported MH mobile application (CS PTSD Coach) to be administered among the WTC GRs.

Florida Sub-Cohort. Florida has seen a significant influx of WTC responders, with over 5,496 registered members. This group is older, more frequently retired, and includes a higher proportion of Latinx individuals compared to responders in other regions. The study focuses on this sub-cohort due to their unique vulnerabilities, including exposure to extreme climate events like hurricanes, which can exacerbate PTSD symptoms. The relocation of WTC responders to Florida is part of a broader trend of population migration from the New York Metropolitan Area to Florida. This trend has resulted in an increasing number of WTCHP members residing in Florida, creating an urgent need for accessible MH services in this region.

Preliminary data indicate that the Florida WTC responders have a high prevalence of PTSD, with an estimated 40% showing probable PTSD symptoms. Additionally, there is a strong interest among these responders in participating in remote-delivered MH services, highlighting the feasibility of the proposed intervention. The data also show that the Florida sub-cohort is older, more frequently retired, and includes a higher proportion of Latinx individuals compared to the overall WTC cohort. The older age of retired GRs, with a higher proportion of Latinx individuals compared to the overall WTC cohort, make the Florida sub-cohort particularly relevant for studying the long-term MH effects of the 9/11 exposures and the potential overlapping impact of aging.

Clinician Supported PTSD Coach Mobile App. The Clinician Supported (CS) PTSD Coach combines self-managed PTSD Coach application with four 20-30 minute psychotherapy sessions delivered by a clinician. The app includes modules on learning about PTSD, self-assessment, symptom management, and finding support. Preliminary studies with veterans have shown that the CS PTSD Coach is effective in reducing PTSD and depression symptoms.

The CS PTSD Coach was originally developed as a brief intervention for Veteran primary care patients with elevated PTSD symptoms who were unlikely to use a mobile app on their own. The intervention combines self-managed PTSD Coach app with four 20-30 minute sessions delivered over eight weeks. These sessions include instructions for app use, setting symptom reduction goals, and assigning PTSD Coach activities for completion between sessions. The clinician sessions help participants select the management strategies within the app that can best address their PTSD symptoms and incorporate these strategies into their daily lives.

PTSD Coach app is available at no cost from iTunes and Google Play marketplaces and is accessible to almost the entire U.S. smartphone-using population. The app is available in both English and Spanish, making it suitable for the diverse population of WTC responders. The primary focus of PTSD Coach is on PTSD symptoms, which include the following: Re-experiencing, intrusive traumatic symptoms such as flashbacks and nightmares; Persistent Avoidance, avoidance of stimuli associated with the traumatic event; Negative Thoughts or Feelings, worsened thoughts or feelings after the traumatic event; and Hyperarousal, symptoms such as sleep disturbances, excessive startle reactions, and irritable behavior. The app provides psychoeducation on trauma and PTSD and helps trauma-exposed individuals monitor and manage their symptoms. It offers cognitive-behavioral-based coping tools such as relaxation exercises, calming self-talk, anger management tools, and effective sleep hygiene practices. The app has also been shown to be effective in reducing symptoms of depression and anxiety, which often co-occur with PTSD.

Significance.

The study is significant for several reasons:

1. Addressing Treatment Gaps: It responds to the need for research on MH interventions for WTC responders, as recommended by the WTCHP Scientific Technical Advisory Committee. The committee has emphasized the importance of further research on MH intervention studies and the effectiveness and utility of PTSD treatments.
2. Focus on Spanish-speaking Latinx Responders: By including this demographic, the study aims to advance health equity. Spanish-speaking Latinx responders have been underrepresented in previous studies, and this research seeks to address their specific needs.
3. Remote Intervention: The use of a mobile application for MH treatment is innovative and necessary for the geographically dispersed WTC responders, especially those in Florida. The app-based intervention provides a scalable and accessible solution to deliver MH care to a large number of responders who may face barriers to accessing traditional in-person treatments.

SPECIFIC AIMS. This study aims to assess the feasibility, acceptability, and efficacy of the PTSD Coach app among a multi-ethnic group of 9/11 GRs in Florida, with a focus on two different versions of the app: clinician-supported (CS) and self-managed (SM). The study includes four aims. The first aim focuses on evaluating engagement levels with the app, analyzing usage data to determine the frequency and duration of interactions, as well as identifying the app modules with the highest engagement across different language groups (English and Spanish). Additionally, feedback on usability, potential barriers, and improvement suggestions will be gathered.

The second aim seeks to evaluate the app's acceptability by examining user satisfaction and using specific measures to gauge positive responses from participants. Feedback on treatment acceptability and appropriateness will also be collected.

The third aim assesses the efficacy of the CS and SM versions of PTSD Coach through a randomized controlled trial (RCT). The primary outcome is the reduction in PTSD symptoms, while secondary outcomes include reductions in depression, anxiety, and sleep disturbances. The study will compare the CS and SM groups with a wait-list control group to evaluate symptom changes post-intervention and follow-up. Additionally, it will investigate whether the CS version is more effective than the SM version and explore potential moderators and mediators of treatment effects.

The final aim focuses on developing and delivering a Spanish-language version of CS PTSD Coach, ensuring that it is feasible, acceptable, and effective for Spanish-speaking participants.

METHODS. Study Design. The study is a two-year project involving a three-arm randomized clinical trial (RCT) with the following three conditions: (1) CS PTSD Coach where participants receive the intervention with clinician support, focusing on app use, symptom monitoring, and management strategies; (2) SM PTSD Coach where participants receive basic instructions on using the app but no further clinician support; and (3) Wait-list Control where participants receive no intervention until after the follow-up assessment when they have a choice of receiving either CS PTSD Coach or SM PTSD Coach. Participants will be assessed at baseline, immediately post-intervention at four weeks, and four weeks later after the intervention. The study aims to evaluate the feasibility, acceptability, and efficacy of PTSD Coach in reducing MH symptoms among WTC responders.

Recruitment and Randomization. Recruitment will leverage existing networks and data from the WTCHP General Responders Data Center. Participants will be randomly assigned to one of the three conditions using a random number generator. The study aims to enroll 120 participants, with a rolling enrollment strategy to ensure sufficient sample size.

Measures and Data Collection. The study uses validated measures to assess PTSD, depression, anxiety, and sleep disturbance symptoms. Data will be collected at multiple time points to evaluate changes in symptoms and the overall effectiveness of the intervention.

Analyses. Continuous data will be summarized using means and standard deviations for normally distributed data. For continuous data that are skewed, medians and interquartile ranges (IQR) will be used to provide a more accurate representation of the central tendency and variability. Categorical data (including binary data) will be summarized using frequency (N) and percent (%). To assess feasibility, acceptability, and efficacy of the interventions, we will employ different approaches to the analyses.

To assess feasibility of PTSD Coach, we will use objective app-use data to first quantify the frequency and duration of interactions with the app and its features. Second, we will analyze usage patterns in these data for peak engagement times and frequency trends in each group, by language. Third, we will identify the specific app modules with the highest engagement rates for the GRs in each group, by language. We will also use the SUS and examine the data to determine if "good" usability is achieved, as noted in the measures section.

To assess acceptability, we will analyze responder satisfaction with PTSD Coach, in both conditions, by language, using the CSQ. Individual items rated as "good" or "excellent" on the CSQ will indicate endorsement by participants. We will also gather feedback about the acceptability of CS PTSD Coach by language group using the AIM and IAM. Items rated as "agree" or "completely agree" will be considered endorsement by participants.

To determine efficacy of CS PTSD Coach, several analyses will be utilized. Paired t-tests will be employed to test changes in psychological symptoms before and after treatment within each condition. This analysis will involve reporting the pre- and post-intervention means and standard deviations to illustrate the extent of change in symptoms. Analysis of Covariance (ANCOVA) will be used to compare changes in symptom scores between the different conditions, CS PTSD Coach, SM PTSD Coach, and the wait-list control. ANCOVA will adjust for baseline scores and other covariates to increase statistical power. Sample size calculations indicate that having 40 participants per group, accounting for a 10% attrition rate, will achieve 80% power to detect significant differences between the conditions.

An intent-to-treat analysis will be conducted, including all participants in the analysis regardless of whether they completed the intervention. To handle missing data, multiple imputation techniques will be used, ensuring that the analysis remains robust and unbiased.

Finally, moderation and mediation analyses will be conducted to further understand the effects of the interventions. Moderators such as baseline PTSD severity, sex, race, ethnicity, and language (English and Spanish) will be examined using interaction terms in the ANCOVA model. Mediation analysis will follow the Baron & Kenny method, utilizing the product-of-coefficient test to assess whether the intervention effect on PTSD symptoms is mediated by other variables.

EXPECTED IMPACT AND CONCLUSION. The study aims to fill critical gaps in MH treatment research for WTC responders, particularly those in Florida. By focusing on a remote, clinician-supported intervention, the study has the potential to improve access to MH care for a geographically dispersed and ethnically diverse population. The findings could inform future research and clinical practice, ultimately enhancing the well-being of WTC responders.

This study represents a significant step forward in addressing the MH needs of WTC responders. By leveraging innovative technology and focusing on an underserved population, it aims to provide effective, accessible, and equitable MH care. The results will have important implications for the broader WTCHP cohort and contribute to the ongoing efforts to support those affected by the 9/11 attacks.

ELIGIBILITY:
Inclusion Criteria:

* World Trade Center General Responders (GRs) currently living in Florida.
* Any age.
* Must have a smartphone device capable of using the PTSD Coach app.
* Must be fluent in either English or Spanish.

Exclusion Criteria:

* Active or recent (past month) suicidal ideation or attempt.
* Low levels of distress as measured by the PCL-5 (score below 30).
* Severe alcohol use measured by an AUDIT score of 20 or above.
* Use of illicit or unprescribed drugs (except for cannabis) in the last 2 weeks, as indicated on the Modified ASSIST Measure.
* Presence of neurologic or neurodegenerative conditions associated with significant cognitive impairment (e.g., Parkinson's, Alzheimer's diseases) or current severe cognitive impairment measured using the Montreal Cognitive Assessment (MoCA).
* Current mental health treatment for PTSD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Evaluate changes in PTSD symptoms from pretest to posttest (8 weeks) and follow-up four weeks later (12 weeks).
  A self-report measure used to assess the presence and severity of PTSD symptoms. It consists of 20 items that correspond to the DSM-5 criteria for PTSD.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9). | Evaluate changes in depression symptoms from pretest to posttest (8 weeks) and follow-up four weeks later (12 weeks).
  Self-report measure that consists of 9 items. Each item corresponds to one of the DSM-5 criteria for depression and is rated on a scale from 0 (not at all) to 3 (nearly every day), based on how often the respondent has been bothered by that symptom over the past two weeks.
Generalized Anxiety Disorder-7 (GAD-7) | Evaluate changes in anxiety symptoms from pretest to posttest (8 weeks) and follow-up four weeks later (12 weeks).
  self-report questionnaire that consists of 7 items, each corresponding to a symptom of generalized anxiety disorder. Respondents rate how often they have been bothered by each symptom over the past two weeks on a scale from 0 (not at all) to 3 (nearly every day)
Insomnia Severity Index (ISI) | Evaluate changes in sleep disturbance symptoms from pretest to posttest (8 weeks) and follow-up four weeks later (12 weeks).
  7-item self-report questionnaire that evaluates the severity of insomnia symptoms over the past two weeks. Each item is rated on a scale from 0 (no problem) to 4 (very severe problem)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Macgowan, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Protecting the privacy of these World Trade Center General Responders is paramount. Sharing IPD could risk exposing sensitive personal information, even if anonymized, which might lead to re-identification.

REFERENCES:
- See also: URL to reference list informing the study protocol — https://drive.google.com/file/d/1udIZ39SgXOy4h9D2SlU0gUwpPEXETHgn/view?usp=sharing